CLINICAL TRIAL: NCT02577952
Title: Lipodystrophy Connect Patient Registry
Status: Completed | Type: Observational
Sponsor: PatientCrossroads (Industry)
Responsible Party: Principal Investigator, Vanessa Rangel Miller, Advocacy Partnerships, PatientCrossroads
Other Study IDs: Pro00009092
Record Dates: First submitted 2015-10-08; First posted 2015-10-16 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Lipodystrophy
Keywords: lipodystrophy; lipodystrophy, congenital generalized; Berardinelli-Seip Congenital Lipodystrophy; Congenital generalized lipodystrophy; generalized lipodystrophy; lipodystrophy, familial partial; partial lipodystrophy; lipodystrophy, partial, acquired; acquired lipodystrophy
MeSH Terms: conditions — Lipodystrophy; Lipodystrophy, Congenital Generalized; Lipodystrophy, Familial Partial; Lipodystrophy, Partial, Acquired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- People with Lipodystrophy & family: People currently living with lipodystrophy and their family members.

SUMMARY:
Lipodystrophy Connect is an online survey tool designed to collect demographic data and health information from individuals with Lipodystrophy.

DETAILED DESCRIPTION:
Lipodystrophy is a heterogeneous group of rare and inherited syndromes characterized by the complete or partial loss or absence of subcutaneous adipose tissue. People living with lipodystrophy lack the fat tissue required for normal metabolic function. To enhance knowledge of the underlying biology of these conditions and to institute effective clinical treatments, the Lipodystrophy community has developed a mechanism for individuals with any of the Lipodystrophy conditions to enroll in a Lipodystrophy registry called Lipodystrophy Connect. The objective of such a registry is to create a platform that connects all of the Lipodystrophy community, including persons with Lipodystrophy, family members, healthcare providers, researchers, drug companies, advocacy groups, federal research organizations, and regulators. A patient registry will provide the foundation for a resource to meet the current and future needs of the Lipodystrophy community as well as accelerate the rate of research and development of therapies that improve the quality of life of those with Lipodystrophy. Lipodystrophy Connect is an online survey tool that collects basic demographic information and health information from people with any rare form of Lipodystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Adults, > 18 years of age, with a diagnosis or suspected diagnosis of lipodystrophy, who are willing and able to provide informed consent, or for whom a legally authorized representative gives permission on behalf of the person to participate.
* Minors (less than 18 years of age) with a diagnosis of lipodystrophy with a parent(s) or legally authorized representative who provides informed consent to participate and enter registry information on behalf of the minor. Note: Minors who are 7-17 years of age will be asked to provide assent to participate.
* Adults > 18 years of age, without lipodystrophy, who are willing and able to provide informed consent and are family members of patients diagnosed with familial partial lipodystrophy (FPL) or congenital generalized lipodystrophy (CGL) and want to provide information about themselves.

Exclusion Criteria:

* A person who does not have a suspected or confirmed diagnosis of Lipodystrophy.
* A person who has a known diagnosis of HIV-associated Lipodystrophy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with known or suspected lipodystrophy and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2014-01; Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Descriptive epidemiology of congenital and acquired lipodystrophy. | Participants are requested to update their questionnaires every 12 months for 5 years.
  Assessed from multiple questions regarding the natural history of patients with congenital or acquired lipodystrophy, with an emphasis on co-morbidities, history of medical evaluation or admission, and use of medications/alternative therapies.

SECONDARY OUTCOMES:
Data on disease subtype | Participants are requested to update their questionnaires every 12 months for 5 years.
  Multiple questions about the patient's diagnostic process including reported diagnosis and subtype, time to diagnosis, method of diagnosis, age at diagnosis, presenting symptoms and specialty of diagnosing clinician.
Change in congenital and acquired lipodystrophy clinical features | Participants are requested to update their questionnaires every 12 months for 5 years.
  Assessed from multiple questions regarding the common physical features hallmark to congenital and acquired lipodystrophy.
Change in patient self-report Quality of Life | Participants are requested to update their questionnaires every 12 months for 5 years.
  Assessed from self-report quality-of-life (QoL) questions about the patient's overall health, everyday living, recent impact, personal impact, available resources, diet and lifestyle history.
Data on family and reproductive history | Participants are requested to update their questionnaires every 12 months for 5 years.
  Multiple questions regarding whether biological family members have been diagnosed with lipodystrophy or report lipodystrophy symptoms, and personal reproductive history.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Rangel Miller, M.S., M.B.A, Principal Investigator — PatientCrossroads
Locations (1):
- PatientCrossroads, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified aggregate participant data is shared via a professional portal.